CLINICAL TRIAL: NCT05952830
Title: Comparison of the Effects of Extracorporeal Shock Wave Therapy and Dry Needing on Spasticity in Poststroke Patients: a Randomized Controlled Trial
Brief Title: Comparison of the Effects of Extracorporeal Shock Wave Therapy and Dry Needing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Buket Büyükturan, associate professor, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 560
Record Dates: First submitted 2023-07-06; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Hemiplegia
Keywords: Hemiplegia; external corporeal shockwave therapy; dry needling; spasticity
MeSH Terms: conditions — Hemiplegia; Muscle Spasticity

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESWT Group (Active Comparator): ESWT Group: external corporeal shockwave therapy subjects in ESWT-group receiving one session shock wave therapy given 6,000 impulses at 0.06-0.07 mJ/mm2 (1.2-1.4 bar) at 18 Hz on biceps brachii
  Interventions: Other: ESWT group
- DN Group (Experimental): DN Group: dry needling Subjects in DN-group receiving dry needling using disposable stain less steel sterilized needles, 0.25×0.30. DN perform with patients in supine position, arm away from the trunk, and forearm in supination. The fast-in and fast-out cone shape technique adopt and each muscle needled for one minute
  Interventions: Other: ESWT group; Other: DN group

INTERVENTIONS:
Other: ESWT group — subjects in ESWT-group receiving one session shock wave therapy given 6,000 impulses at 0.06-0.07 mJ/mm2 (1.2-1.4 bar) at 18 Hz on biceps brachii (17). Subjects in DN-group receiving dry needling using disposable stain less steel sterilized needles, 0.25×0.30. DN perform with patients in supine position, arm away from the trunk, and forearm in supination. The fast-in and fast-out cone shape technique adopt and each muscle needled for one minute
Other: DN group — Subjects in DN-group receiving dry needling using disposable stain less steel sterilized needles, 0.25×0.30. DN perform with patients in supine position, arm away from the trunk, and forearm in supination. The fast-in and fast-out cone shape technique adopt and each muscle needled for one minute
  Arms: DN Group

SUMMARY:
Effective treatment of spasticity after stroke is a very important and serious problem. Some of the therapeutic approach include physiotherapy and medication. In the recent years external corporeal shockwave therapy and dry needling are commonly used for management of spasticity and pain after stroke. the purpose of this study is the comparative study between effectiveness of external corporeal shockwave therapy (ESWT) and dry needling (DN) on spasticity, pain, and upper limb function and sensation in individuals with hemiplegia.

Methods: In this study, individuals with hemiplegia were randomized 1:1 to parallel ESWT-Group (n = 10) or DN group (CG) (n = 10). Upper Extremity Functions, Sensation, Spasticity and Pain were evaluated. All measurement indicators were be evaluate before treatment and immediately after one session treatment. Mixedmodel repeated measured ANOVAs were then employed to determine if a group*time interaction existed on the effects of the treatment on each outcome variable for each group as the between-subjects variable and time as the within-subjects variables.

DETAILED DESCRIPTION:
Effective treatment of spasticity after stroke is a very important and serious problem. Some of the therapeutic approach include physiotherapy and medication. In the recent years external corporeal shockwave therapy and dry needling are commonly used for management of spasticity and pain after stroke. the purpose of this study is the comparative study between effectiveness of external corporeal shockwave therapy (ESWT) and dry needling (DN) on spasticity, pain, and upper limb function and sensation in individuals with hemiplegia.

Methods: In this study, individuals with hemiplegia were randomized 1:1 to parallel ESWT-Group (n = 10) or DN group (CG) (n = 10). Upper Extremity Functions, Sensation, Spasticity and Pain were evaluated. All measurement indicators were be evaluate before treatment and immediately after one session treatment. Mixedmodel repeated measured ANOVAs were then employed to determine if a group*time interaction existed on the effects of the treatment on each outcome variable for each group as the between-subjects variable and time as the within-subjects variables.

ELIGIBILITY:
Inclusion Criteria:

* being between the age of 25-65
* having been diagnosed with a stroke by a specialist, first time stroke
* BBM spasticity, ability to understand command actions
* stable vital signs, unchanged drug doses that might affect muscle spasticity
* taking no antispastic medication
* with Modified Ashworth Scale (MAS) score more than 1 and less than 4 for the upper limb flexor tension

Exclusion Criteria:

* received Botox, alcohol or phenol block treatments
* received elbow joint surgical orthopedic surgery
* history of epilepsy
* severe mental disorders
* malignant tumors; and limb venous thrombosis
* sensory disturbances
* the presence of any other neurological disorders
* currently receiving other treatments
* ESWT contraindications
* exhibit fear of needles; or have any contraindication to DN

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-08-21 (Actual); Primary Completion 2021-08-21 (Actual); Study Completion 2021-10-26 (Actual)

PRIMARY OUTCOMES:
Jebsen Taylor Test of Hand Function (JTHF) | 1 month
  To do JTHF the participant seat on a chair in front of a table. The test consist of 7 parts. For the first part (writing) individuals will be given a blank A4 paper and a pen and asked to write a sentence shown to them. For the second part (page turning task), a booklet with A4 paper size pages will be given to the individual and asked to turn 5 pages as fast as possible. For the third part (collecting and dropping small objects), 2 covers, 2 book clips and 2 coins will be used. These materials will be placed on a plate, spaced apart, on the table, right in front of the individual's hand to administer the test.
Purdue Pegboard Test (PPT) | 1 month
  : To do PPT, the participant seat on a chair in front of a table while the board is on the table. Nails a washers placed in the holes above the board. After the explanation of the test and letting the participant to practice; the test starts. The patient must put the nails in 30 second in the first 3 test; the maximum number that he or she can is the test result. first with the non affected hand, then with the other hand, and finally with both hands simultaneously from top to bottom. In the final subtest, individuals will use both hands to construct sets of nails and washers in a 60-second period. Finally, the combining score consists of the number of sets of nails and stamps collected (22,23).
9 Hole Peg Test | 1 month
  To do 9 hole peg test (9-HPT), the participant seat on a chair in front of a table while the board is on the table. the sticks are on the affected hand side of the individuals and the holes are on the non-affected hand side. The participants must place the sticks in holes and then remove them from the holes as quickly as possible After the explanation of the test and letting the participant to practice; the test starts. Test results will be recorded by measuring the time with a stopwatch from the moment individuals touch the first stick until the last stick is inserted into the board (21).
Spasticity | 10 minutes
  We used modified ashworth scale to test spasticity in elbow flexors while the participants lying supine.

SECONDARY OUTCOMES:
Light Touch | 1 month
  In light touch test we used a cotton swab to touth each area include arm, forearm, hand and finger. İn each test we asked the patient to sey yes or no if he/she could sense the swab while the patiant is in a supine position, upper limb at the side with eyes closed. If there is no loss of light touch feeling, "0 point" will be given, if there is, "1 point" will be given. Then for total grading the grade of each area sum together
Tactile Sense | 1 month
  Patient in a supine position, upper limb at the side and eyes closed. At the first step we start with thickest filament (6.65) and we pressed against the skin at a 90º angle until it begins to bend to half its length, then we asked the patient if he or she could sense the filament or not. If the patient could sense this filament we test the another filament with less thickness (5.58). this process continue until the patient couldn't sense a filament. The first value that cannot be felt from the applied filament thickness values will be recorded. This test performed in arm, forearm, hand and finger (25).
Pain Sensation | 1 month
  For pain sensation test the patient must be in supine position, upper limb at the side with closed eyes. Then we used a discriminator with sharp and blunt head. We randomly alternating sharp or blunt pressure. We asked the patient to response blunt if he/she sense "blunt" and response "sharp" if he/she sense sharp. We examined this test in arm, forearm, hand and finger. If there is no loss in the sense of pain, "0 point" will be given, if there is, "1 point" will be given. Then for total grading the grade of each area sum together
2 Point Discrimination | 1 month
  : For 2 point discrimination (2PD) the patient was in a supine in supine position, upper limb at the side with closed eyes. At the first step examiner use the widest discriminator gap [100 millimeters (mm)]. The we asked the patiant to saide if he/she sense one point or two point. İf the patiant felt one point the test stop but if she could sense 2 point we decrease the distence and then aske again. This prosses continue and the decrease the distance and eventually to the narrowest gap (1mm). the narrowest gap felt as a single point will be recorded as the measurement value. We examined this test in arm, forearm, hand and finger.
Visual Anolog Scale | 1 month
  We used Visual Anolog Scale (VAS) to assessed pain. We completed the VAS before and immediately after one session of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hüseyin Abdul Razzaq Cabbar Sarefi, PT, Study Director — Karbala Health Department.
Locations (2):
- Turkey (Türkiye) (2):
  - Ahi Evran University, Kırşehir, Merkez
  - Kırşehir Ahi Evran University, Kırşehir, Merkez